CLINICAL TRIAL: NCT00395460
Title: A Single-blind, Multicenter, Randomized, Phase III Study of the Efficacy and Safety of Gadavist (1.0 M) in Comparison With Magnevist (0.5 M) as Contrast Agent for Enhanced Magnetic Resonance Imaging (MRI) of Central Nervous System (CNS) Lesions in Chinese Patients
Brief Title: Efficacy and Safety Study to Evaluate Gadavist (Gadobutrol) as Contrast Agent in Magnetic Resonance Imaging (MRI) of Brain or Spine Diseases in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 91536; Project DE 00562 (Other: Company internal); 309761 (Other: Company internal)
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2011-11-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Central Nervous System Diseases
Keywords: Gadovist; Gadavist; Contrast agent; Brain; Spine disease; Magnetic Resonance Imaging
MeSH Terms: conditions — Central Nervous System Diseases; Spinal Diseases | interventions — gadobutrol; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gadobutrol 0.1 mmol/kg Body Weight (BW) (Gadavist, BAY86-4875) (Experimental): Participant received 0.1 mmol/kg BW Gadobutrol (= 0.1 mL/kg BW by intravenous injection at a rate of 1.0 mL/sec)
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- GD 0.1 mmol/kg BW (Magnevist, BAY86-4882) (Active Comparator): Participant received 0.1 mmol/kg BW Gadopentetate Dimeglumine (GD) (= 0.2 mL/kg BW by intravenous injection at a rate of 2.0 mL/sec
  Interventions: Drug: Magnevist

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — 1,0M, intra venous injection at a dose of 0,1 ml/kg BW (= 0,1 mmol Gd/kg BW)
  Arms: Gadobutrol 0.1 mmol/kg Body Weight (BW) (Gadavist, BAY86-4875)
Drug: Magnevist — 0,5M, intra venous injection at a dose of 0,2 ml/kg BW (= 0,1 mmol Gd/kg BW)
  Arms: GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)

SUMMARY:
The purpose of this study is to determine if the contrast agent is effective and safe in the Magnetic Resonance Imaging (MRI) of brain or spine diseases in patients of Chinese origin.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin, with known or suspected brain or spine diseases

Exclusion Criteria:

* Pregnancy
* Lactation
* Conditions interfering with MRI
* Allergy to any contrast agent or any drugs
* Participation in other trial
* Require emergency treatment
* Severely impaired liver and kidney functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- China (4):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The 1st Affiliated Hosp of the 4th Military Med Uni, Xi'an, Shaanxi
  - Chinese PLA General Hosp., Beijing
  - Fudan University Huashan Hospital, Shanghai

REFERENCES:
- [Result] Liang Z; Ma L; Wang D; Huan Y; Li P; Yu J; Yao Z; Chen S; He H; Feng X and Breuer J. Efficacy and Safety of Gadobutrol (1.0 M) versus Gadopentetate Dimeglumine (0.5 M) for Enhanced MRI of CNS Lesions: A Phase III, Multicenter, SingleBlind, Randomized Study in Chinese Patients. Magnetic Resonance Insights 2012; 5:17-28

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at specialized study centers if they satisfied the inclusion and exclusion criteria. All had known or suspected central nervous system lesions (including cranial and spinal lesions) with an indication for contrast enhanced magnetic resonance imaging for diagnosis and further treatment.
Pre-assignment Details: Of 150 screened participants, 3 were not randomized (2 due to withdrawal of consent, and 1 due to poor physical condition). 147 participants were randomized to either Gadobutrol 0.1 mmol/kg body weight (BW) (72 participants) or Gadopentetate dimeglumine 0.1 mmol/kg BW (75 participants).
Groups:
- Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875): Participant received 0.1 mmol/kg BW Gadobutrol (= 0.1 mL/kg BW by intravenous injection at a rate of 1.0 mL/sec)
Period: Overall Study
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Started | 72 | 75
Received Treatment | 71 (1 participant withdrew consent prior to study drug injection and did not receive any study drug.) | 75
Completed | 71 | 75
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882) | Total
Number analyzed (Participants) | 71 | 75 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.24) | 43.9 (10.1) | 43.4 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 75
  Male | 38 | 33 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Contrast to Noise Ratio (CNR) Between Pre- and Post-contrast Magnetic Resonance Imaging (MRI) Scan of Central Nervous System (CNS) Lesions
Description: CNR = (signal intensity [SI] lesion - SI normal tissue) / standard deviation (SD) background. SI lesion is the signal intensity in the lesion, SI normal tissue is the signal intensity in the normal tissue, and SD background is the standard deviation of the background noise. The signal intensity (SI) on the pre-contrast and on the post-contrast MR scans was to be measured in the enhanced lesion, normal tissue and background.
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases. Two participants in each treatment group had missing values for signal intensity for central nervous system lesions at pre- and post-contrast and could thus not be considered for evaluation.
Measure: Mean (Standard Deviation); unit: Contrast to Noise ratio
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 68 | 73
Contrast to Noise ratio | 50.41 (38.448) | 43.47 (39.178)
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) vs GD 0.1 mmol/kg BW (Magnevist, BAY86-4882); Test type: Non-Inferiority or Equivalence — The analysis was performed by means of a Confidence Interval (CI) approach: noninferiority of Gadavist was assumed if the one-sided 95% CI for pGadavist-pMagnevist was lying entirely to the right of the value -delta, where p is the estimated change in CNR and with pre-defined non-inferiority margin delta of 15% (=6.52 or 15% of 43.467); non-inferiority; Mean Difference (Final Values) = 6.939, 95% CI 1-sided [lower limit -3.897], Standard Deviation 38.83

2. Secondary Outcome: Change in Number of Detected Lesions From Pre- to Post-contrast MRI Scan
Description: The number of lesions in the magnetic resonance scans was recorded before and after injection of contrast agent for the investigators and all 3 blinded readers (reader 2, reader 3 and reader 4).
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 70 | 75
Lesions
  Investigator | 0.7 (2.56) | 0.1 (0.83)
  Reader 2 | 1.4 (6.94) | 0.3 (1.87)
  Reader 3 | 1.7 (9.72) | 0.3 (1.44)
  Reader 4 | 0.5 (2.72) | 0.1 (0.93)

3. Secondary Outcome: Change in Diagnostic Confidence From Pre- to Post-contrast Magnetic Resonance Imaging by Treatment
Description: The change in diagnostic confidence was assessed based on post-contrast compared to pre-contrast scans as "improved", "unchanged" or "worsened" for the investigators and all 3 blinded readers (reader 2, reader 3 and reader 4).
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases.
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 70 | 75
Participants
  Investigator - improved | 68 | 65
  Investigator - unchanged | 2 | 10
  Investigator - worsened | 0 | 0
  Reader 2 - improved | 55 | 61
  Reader 2 - unchanged | 15 | 14
  Reader 2 - worsened | 0 | 0
  Reader 3 - improved | 59 | 61
  Reader 3 - unchanged | 11 | 14
  Reader 3 - worsened | 0 | 0
  Reader 4 - improved | 60 | 63
  Reader 4 - unchanged | 8 | 12
  Reader 4 - worsened | 2 | 0

4. Secondary Outcome: Change in Lesion Contrast Enhancement From Pre- to Post-contrast MRI
Description: The degree of contrast enhancement was recorded on a 4-point scale as follows: 1 = No: lesion is not enhanced. 2 = Moderate: lesion is weakly enhanced. 3 = Good: lesion is clearly enhanced. 4 = Excellent: lesion is clearly and brightly enhanced. In case of more than one lesion, the lesion with maximum enhancement was to be assessed. The change in lesion contrast enhancement was assessed based on post-contrast in comparison to pre-contrast scans for the investigators and all 3 blinded readers (reader 2, reader 3 and reader 4).
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases. Lesion contrast enhancement of 1 participant in the Gadavist group was assessed by the investigator (but not the blinded readers) as 'not applicable'.
Measure: Mean (Standard Deviation); unit: Contrast enhancement score
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 70 | 75
Contrast enhancement score
  Investigator | 2.4 (0.87) | 2.2 (0.87)
  Reader 2 | 2.1 (1.21) | 2.0 (1.22)
  Reader 3 | 1.7 (0.98) | 1.6 (0.89)
  Reader 4 | 2.2 (1.05) | 2.1 (1.09)

5. Secondary Outcome: Change in Lesion Delineation Between Pre- and Post-contrast MRI Scan of CNS Lesions
Description: Lesion delineation was recorded on a 4-point scale as follows: 1 = None: no or unclear delineation of the boundary between lesion and surrounding tissue; 2 = Moderate: some aspects of border delineation covered; 3 = Good: almost clear delineation, but not complete on relevant slices; 4 = Excellent: sharp and complete delineation. In case of more than one lesion, the lesion with maximum enhancement was assessed. Change in lesion delineation was assessed based on post-contrast in comparison to pre-contrast scans for investigators and all 3 blinded readers (reader 2, reader 3 and reader 4).
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Lesion delineation score
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 70 | 75
Lesion delineation score
  Investigator | 1.1 (0.73) | 1.0 (0.85)
  Reader 2 | 1.4 (0.89) | 1.3 (0.88)
  Reader 3 | 0.9 (0.71) | 0.8 (0.53)
  Reader 4 | 1.0 (0.81) | 0.9 (0.67)

6. Other Pre Specified Outcome: Change in Contrast to Noise Ratio (CNR) Between Pre- and Post-contrast MRI Scan of CNS Lesions in Participants With Malignant Brain Tumor(s) / Brain Metastases
Description: CNR = (SI lesion - SI normal tissue) / SD background. SI lesion is the signal intensity in the lesion, SI normal tissue is the signal intensity in the normal tissue, and SD background is the standard deviation of the background noise. The signal intensity (SI) on the pre-contrast and on the post-contrast MR scans was to be measured in the enhanced lesion, normal tissue and background.
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All valid case participants who received contrast injection. Subgroup: those with primary malignant brain tumor(s) / brain metastases. One participant in the Gadavist group had missing values for signal intensity for central nervous system lesions at pre- and post-contrast and could thus not be considered for evaluation.
Measure: Mean (Standard Deviation); unit: Contrast to Noise ratio
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 20 | 25
Contrast to Noise ratio | 54.95 (42.405) | 46.56 (30.074)

7. Other Pre Specified Outcome: Change in Contrast to Noise Ratio (CNR) Between Pre- and Post-contrast MRI Scan of Participants With CNS Lesions Other Than Primary Malignant Brain Tumor(s) / Brain Metastases
Description: as for outcome 6
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All valid case participants who received contrast injection. Subgroup: those with CNS lesions other than primary malignant brain tumor(s) / brain metastases. 1 (Gadavist) and 2 participants (Magnevist) had missing values for signal intensity for CNS lesions pre- and post-contrast and could not be considered for evaluation.
Measure: Mean (Standard Deviation); unit: Contrast to Noise ratio
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 48 | 48
Contrast to Noise ratio | 48.51 (36.985) | 41.86 (43.379)

8. Other Pre Specified Outcome: Change in Number of Detected Lesions From Pre- to Post-contrast MRI Scan of CNS Lesions in Participants With Malignant Brain Tumor(s) / Brain Metastases
Description: Investigators and blinded readers (reader 2, 3 and 4) were to record the number of lesions in the magnetic resonance scans before and after injection of contrast agent.
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases. Subgroup: participants with primary malignant brain tumor(s) / brain metastases
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 21 | 25
Lesions
  Investigator | 0.7 (2.61) | 0.4 (1.41)
  Reader 2 | 0.4 (1.75) | 0.2 (0.55)
  Reader 3 | 0.5 (2.18) | 0.2 (0.72)
  Reader 4 | 0.1 (0.30) | 0.0 (0.20)

9. Other Pre Specified Outcome: Change in Number of Detected Lesions From Pre- to Post-contrast MRI Scan of Participants With CNS Lesions Other Than Primary Malignant Brain Tumor(s) / Brain Metastases
Description: Investigators and blinded readers (reader 2, 3 and 4= were to record the number of lesions in the magnetic resonance scans before and after injection of contrast agent.
Time Frame: Immediately before injection (pre-contrast) and 2-5 min after injection (post-contrast)
Population: Per Protocol Set (PPS): All patients who have received contrast injection and are not invalid cases. Subgroup: participants with CNS lesions other than primary malignant brain tumor(s) / brain metastases
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Number analyzed (Participants) | 49 | 50
Lesions
  Investigator | 0.7 (2.57) | 0 (0)
  Reader 2 | 1.8 (8.20) | 0.3 (2.26)
  Reader 3 | 2.2 (11.53) | 0.3 (1.70)
  Reader 4 | 0.7 (3.24) | 0.2 (1.13)

ADVERSE EVENTS:
Arm/Group | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882)
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/75
Other Adverse Events (participants affected / at risk) | 2/71 | 4/75
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) (N=71) | GD 0.1 mmol/kg BW (Magnevist, BAY86-4882) (N=75)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs shall provide sponsor with an advance copy of any proposed publication or oral presentation at least ninety (90) days prior to the date of the planned submission or presentation. Sponsor shall have sixty (60) days to recommend any changes it reasonably believes are necessary for scientific purposes or to preserve the confidentiality of sponsor's confidential information. PIs agree that the adoption of such recommended changes shall not be unreasonably refused.